CLINICAL TRIAL: NCT01297920
Title: A Three-Month, Randomized, Double-Masked, Parallel-Group Study With a Planned Three-Month Safety Extension of the Efficacy and Safety of a Fixed Combination of Brinzolamide 1%/Brimonidine 0.2% Compared to Brinzolamide 1% and Brimonidine 0.2% All Dosed Three Times Daily in Patients With Open-Angle Glaucoma and/or Ocular Hypertension
Brief Title: Three Month Efficacy/Safety Study With a 3-Month Safety Extension of Brinzolamide 1%/Brimonidine 0.2% vs. Brinzolamide 1% or Brimonidine 0.2%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-10-039
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-05

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-Angle Glaucoma; Ocular Hypertension; Brinzolamide; Brimonidine; Intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brinz/Brim (Experimental): Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension, 1 drop instilled in each eye 3 times a day for 3 months
  Interventions: Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension
- Brinzolamide (Active Comparator): Brinzolamide ophthalmic suspension, 1%, 1 drop instilled in each eye 3 times a day for 3 months
  Interventions: Drug: Brinzolamide ophthalmic suspension, 1%
- Brimonidine (Active Comparator): Brimonidine tartrate ophthalmic solution, 0.2%, 1 drop instilled in each eye 3 times a day for 3 months
  Interventions: Drug: Brimonidine tartrate ophthalmic solution, 0.2%

INTERVENTIONS:
Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension
  Arms: Brinz/Brim
Drug: Brinzolamide ophthalmic suspension, 1%
  Arms: Brinzolamide
Drug: Brimonidine tartrate ophthalmic solution, 0.2%
  Arms: Brimonidine

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of a new ophthalmic suspension (Brinz/Brim) in lowering intraocular pressure (IOP) relative to its individual active components in subjects with open-angle glaucoma and/or ocular hypertension.

DETAILED DESCRIPTION:
This study consisted of 7 visits conducted during 2 sequential phases: the screening/eligibility phase, which included a screening visit and 2 eligibility visits, and the treatment phase, which included 4 on-therapy visits conducted at Week 2, Week 6, Month 3, and Month 6. A washout period based on previous ocular medication preceded Eligibility Visit 1. Subjects who met all inclusion/exclusion criteria at both eligibility visits were randomized to 1 of 3 study drug groups. The study was designed to evaluate the efficacy and safety of Brinzolamide/Brimonidine over a 3-month period, with an additional 3 months of study drug exposure intended to provide further safety data.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent document.
* Diagnosis of open-angle glaucoma or ocular hypertension, with mean intraocular pressure within protocol-specified range at eligibility visit/s.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential if pregnant, lactating, or not using highly effective birth control measures.
* Any form of glaucoma other than open-angle glaucoma.
* Severe central vision loss in either eye.
* Chronic, recurrent, or severe inflammatory eye disease.
* Ocular trauma within the preceding 6 months.
* Ocular infection or ocular inflammation within the preceding 3 months.
* Clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy, or retinal detachment.
* Best-corrected visual acuity score worse than 55 letters using the Early Treatment Diabetic Retinopathy Study chart.
* Other ocular pathology (including severe dry eye) that may, in the opinion of the Investigator, preclude the administration of study product.
* Ocular surgery within the preceding 6 months.
* Ocular laser surgery within the preceding 3 months.
* Any abnormality preventing reliable applanation tonometry.
* Any other conditions, including severe illness, which could make the subject, in the opinion of the Investigator, unsuitable for the study.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1062 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Teague, BS, Sr. Clinical Manager, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited and enrolled from 64 investigational centers in the United States.
Pre-assignment Details: Of the 1062 enrolled, 372 subjects did not meet inclusion/exclusion criteria and were exited from the study as screen failures prior to randomization. This reporting group includes all randomized subjects (690), as treated.
Period: Overall Study
Arm/Group | Brinz/Brim | Brinzolamide | Brimonidine
Started | 221 | 234 | 235
Completed | 163 | 207 | 178
Not Completed | 58 | 27 | 57
Not completed — Adverse Event | 42 | 10 | 38
Not completed — Patient Decision Unrelated to AE | 6 | 5 | 2
Not completed — Noncompliance | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 3 | 0
Not completed — Inadequate Control of IOP | 7 | 9 | 17
Not completed — Patient Did Not Meet Entrance Criteria | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized subjects, as treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brinz/Brim | Brinzolamide | Brimonidine | Total
Number analyzed (Participants) | 221 | 234 | 235 | 690
Age, Customized [Number; unit: participants]
  18 to 64 years | 99 | 113 | 115 | 327
  ≥65 years | 122 | 121 | 120 | 363
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 136 | 132 | 387
  Male | 102 | 98 | 103 | 303
Region of Enrollment [Number; unit: participants]
  United States | 221 | 234 | 235 | 690

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure (IOP) at Each Assessment Timepoint (8 AM, +2 h, +7 h, and +9 h) at Month 3
Description: The study drug was instilled at 8 AM and 3 PM (approximately 15 minutes after conducting the IOP measurements). Intraocular pressure was measured by Goldmann applanation tonometry. One eye from each patient was chosen as the study eye and only data for the study eye were used for the efficacy analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Month 3
Population: Intent-to-Treat (ITT): All subjects who received study medication and completed at least 1 scheduled on-therapy study visit. Observed case analysis of the ITT dataset, per randomized treatment assignment.
Measure: Least Squares Mean (Standard Error); unit: millimeters mercury (mm HG)
Arm/Group | Brinz/Brim | Brinzolamide | Brimonidine
Number analyzed (Participants) | 196 | 216 | 203
millimeters mercury (mm HG)
  8 AM (before study drug instillation) | 21.1 (0.30) | 22.0 (0.29) | 23.2 (0.30)
  + 2 hours relative to 8 AM dosing | 18.0 (0.30) | 20.8 (0.29) | 19.9 (0.30)
  + 7 hours relative to 8 AM dosing | 19.5 (0.30) | 20.7 (0.29) | 21.5 (0.30)
  + 9 hours relative to 8 AM dosing | 17.2 (0.30) | 20.4 (0.29) | 18.9 (0.30)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. The safety population includes all subjects who were exposed to study drug.
Description: An adverse event was any untoward medical occurrence in a subject exposed to study drug. The AE did not necessarily have to have had a causal relationship with the study drug. Reports of AEs were obtained through solicited and spontaneous comments from the subjects and through observations by the Investigator as outlined in the study protocol.
Arm/Group | Brinz/Brim | Brinzolamide | Brimonidine
Serious Adverse Events (participants affected / at risk) | 7/221 | 7/234 | 7/235
Other Adverse Events (participants affected / at risk) | 53/221 | 35/234 | 27/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brinz/Brim (N=221) | Brinzolamide (N=234) | Brimonidine (N=235)
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Aortic aneurysm repair (Surgical and medical procedures) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Nephrectomy (Surgical and medical procedures) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Prostatectomy (Surgical and medical procedures) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Retinal tear (Eye disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Intervertebral disc operation (Surgical and medical procedures) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Otitis media chronic (Infections and infestations) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brinz/Brim (N=221) | Brinzolamide (N=234) | Brimonidine (N=235)
Conjunctivitis (Eye disorders) | 16 | 0 | 15
Vision blurred (Eye disorders) | 12 | 18 | 1
Eye allergy (Eye disorders) | 14 | 1 | 5
Eye irritation (Eye disorders) | 14 | 6 | 9
Dysgeusia (Nervous system disorders) | 9 | 24 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.